



# Identificação das necessidades dos usuários de próteses em relação aos seus dispositivos

#### Novembro 2023

#### 1. Resumo

Apesar de muitos avanços no desenvolvimento de próteses, ainda há algumas áreas que precisam de ser melhoradas. Uma delas é o peso dos dispositivos, que pode causar fadiga muscular no uso prolongado da prótese e até mesmo o seu abandono. Este estudo visa identificar as melhorias desejadas nos dispositivos protésicos na perspetiva dos utilizadores, terapeutas e familiares. Isso seria feito através de dois tipos de questionários sobre a aceitação da tecnologia.

# 2. Definição do problema

A Organização Mundial de Saúde (OMS) estima que cerca de 1,3 mil milhões de pessoas sofrem de deficiências significativas. Um dos desafios actuais é facilitar e quebrar as barreiras das pessoas com deficiência. A tecnologia de assistência auxilia a inclusão e a participação, principalmente de pessoas com deficiência.

No Brasil, o DATASUS estimou que cerca de 57802 amputações (um tipo de deficiência) foram realizadas em 2022. As próteses são dispositivos assistivos que visam amenizar o impacto psicológico da falta de um membro e auxiliar nas atividades da vida diária (AVD). Um tipo de prótese é a eléctrica, que utiliza componentes eléctricos para acionar o dispositivo e é normalmente controlada por sinais corporais, como a eletromiografia de superfície (sEMG). Apesar dos muitos avanços no desenvolvimento de próteses, algumas áreas precisam de ser melhoradas, como o peso, o tamanho, o design ergonômico, etc. dos dispositivos, que podem causar fadiga muscular no uso prolongado da prótese e até mesmo o seu abandono.

#### 3. Justificativa e uso dos resultados

Este estudo tem como objetivo identificar os aspectos que causam maior desconforto nos utilizadores de próteses do membro superior. Além disso, reconhecer em quais atividades da vida diária, a prótese está envolvida. Essas informações serão utilizadas para melhorar o design de uma prótese de membro superior.

# 4. Objetivo

#### 4.1. Objetivo Geral

Este estudo visa identificar as melhorias desejadas nos dispositivos protésicos na perspetiva dos utilizadores, terapeutas e familiares.

#### 4.2. Objetivo Especifico

- Fazer um questionário com os utilizadores amputados
- Elaborar um questionário com os terapeutas





• Elaborar um questionário com os familiares dos utilizadores amputados

## 5. Metodologia

Para a execução, serão utilizados três tipos de questionários sobre a aceitação da tecnologia. No primeiro questionário, destinado aos utilizadores de próteses, haverá 15 questões para identificar que tipo de atividades a pessoa utiliza a prótese, qual o tempo de utilização e qual o principal problema com o dispositivo. No segundo e terceiro questionário, destinado ao terapeuta e familiares respectivamente, haverá entre 8 e 9 perguntas para analisar quais as características do aparelho eles acham que causam maior desconforto nos usuários de prótese durante o uso e que poderiam ser melhoradas.

## 5.1. Tipo de estudo

Estudo observacional, qualitativo-quantitativo

## 5.2. Critérios de elegibilidade

Usuários de próteses com pelo menos 6 meses de utilização do dispositivo. Terapeutas com experiência no trabalho com amputados. Familiares dos utilizadores de próteses que vivem com eles.

## 5.3. Equipamentos e instalações

- Questionários de aceptação da tecnologia para os usuários de prótese.
- Questionários de aceptação da tecnologia para os familiares.
- Questionários de aceptação da tecnologia para os terapeutas.
- Os teste sarão realizados nas instalações do CREFES ou nas instalações da UFES.

#### 5.4. Intervenção proposta

A intervenção proposta é descrita a seguir:

- 1. Familiarização com nosso grupo de pesquisa, explicando o objetivo do estudo.
- 2. Realização dos questionários com os usuários de prótese, os familiares e os terapeutas.

#### 5.5. Obtenção de dados

Para a coleta de dados, será usado um telefone celular em que um dos três questionários feitos no Google Forms será aberto e respondido no mesmo dispositivo com a ajuda do pesquisador. Os dados serão salvos imediatamente no Google Drive.

#### 6. Consentimento informado

O consentimento informado deste protocolo é dirigido a usuários de próteses, familiares e terapeutas que participarão do estudo. A seção é dividida em duas partes principais: as informações sobre o estudo e o formulário de consentimento que o paciente deve assinar e, assim, aceitar que seus dados pessoais sejam usados.





## 6.1. Propósito

A Organização Mundial de Saúde (OMS) estima que cerca de 1,3 mil milhões de pessoas sofrem de deficiências significativas. Um dos desafios actuais é facilitar e quebrar as barreiras das pessoas com deficiência. A tecnologia de assistência auxilia a inclusão e a participação, principalmente de pessoas com deficiência.

No Brasil, o DATASUS estimou que cerca de 57802 amputações (um tipo de deficiência) foram realizadas em 2022. As próteses são dispositivos assistivos que visam amenizar o impacto psicológico da falta de um membro e auxiliar nas atividades da vida diária (AVD). Um tipo de prótese é a eléctrica, que utiliza componentes eléctricos para acionar o dispositivo e é normalmente controlada por sinais corporais, como a eletromiografia de superfície (sEMG). Apesar dos muitos avanços no desenvolvimento de próteses, algumas áreas precisam de ser melhoradas, como o peso, o tamanho, o design ergonômico, etc. dos dispositivos, que podem causar fadiga muscular no uso prolongado da prótese e até mesmo o seu abandono.

Este estudo tem como objetivo identificar os aspectos que causam maior desconforto nos utilizadores de próteses do membro superior. Além disso, reconhecer em quais atividades da vida diária, a prótese está envolvida. Essas informações serão utilizadas para melhorar o design de uma prótese de membro superior.

## 6.2. Tipo de pesquisa

Essa pesquisa inclui um protocolo não invasivo, todos os testes serão realizados por um ou dois membros do grupo de pesquisa que está desenvolvendo o projeto.

#### 6.3. Critérios de elegibilidade

Usuários que tenham sido previamente selecionados por meio do protocolo de seleção de pacientes; esses pacientes devem concordar com os testes a serem realizados.

## 6.4. Procedimento y protocolos

No processo desse protocolo, serão considerados 30 participantes amputados, 30 membros da família e 10 terapeutas, cada um dos quais preencherá um questionário com a ajuda de pelo menos um membro do grupo de pesquisa. O tempo entre a familiarização e o preenchimento do questionário é estimado em 60 minutos.

- 1. Familiarização com nosso grupo de pesquisa, explicando o objetivo do estudo.
- 2. Realização dos questionários com os usuários de prótese, os familiares e os terapeutas.

#### 6.5. Metodologia

Você não é obrigado a participar desta pesquisa se não quiser. Você pode deixar a pesquisa a qualquer momento. Todos os seus direitos serão sempre respeitados.

#### 6.6. Benefícios e desconfortos

Sua participação neste estudo contribui para o progresso da pesquisa e talvez no futuro mais pessoas possam se beneficiar de sua participação. Você não sentirá nenhum desconforto durante este estudo.

#### 6.7. Incentivos

Nenhum incentivo será dado por fazer parte da pesquisa.

#### 6.8. Confidencialidade

Todas as informações obtidas nesses testes serão registradas e armazenadas de forma anônima, ou seja, seu nome e seus dados pessoais nunca serão divulgados ou publicados.





## 6.9. Compartimento dos resultados

Durante o estudo, os participantes poderão se informar sobre o status e os resultados preliminares do projeto. Os resultados finais da pesquisa serão tornados públicos para que outras pessoas interessadas possam conhecê-los e ter acesso a eles. Nenhuma informação confidencial será compartilhada.

| 6.10. Consentime | ento informado |
|---|---|
| Eu, | , identificado com o CPF |
| mente; portanto, dou me<br>necessidades dos usuário | ndi o presente documento e que minhas perguntas foram respondidas satisfatoria u consentimento informado para participar da pesquisa intitulada Ïdentificação da s de próteses em relação aos seus dispositivos". Concordo que meu nome, idadenétricos sejam armazenados. Sei que posso me retirar do experimento a qualque |
| Dados do participant | 2 |
| Endereço | |
| Teléfone | |
| Assinatura | CPF |
| Declaração do pesqui | sador |
| de sua participação e os p | i a esta pessoa a natureza e o objetivo da pesquisa, e que ela compreende a natureza<br>cossíveis riscos e benefícios envolvidos. Todas as perguntas que essa pessoa fez foran<br>nte. Também li e expliquei adequadamente as partes do formulário de consentimento |
| informado. Afirmo, por i | neio de minha assinatura. |
| Pesquisador | |
| Assinatura | CPF |

# 7. Questionários

## 7.1. Questionário usuário de prótese

- 1. Gênero
  - Feminino
  - Masculino
  - Não Binário
  - Prefere n\u00e3o responder
- 2. Idade
  - **18-20**
  - **21-30**
  - **31-40**
  - **41-50**
  - **51-60**
- 3. Nível da amputação
  - Ombro
  - Cotovelo
  - Pulso



4. Tipo de prótese que usa

# Universidade Federal do Espírito Santo Identificar as necessidades dos usuários de próteses em relação aos seus dispositivos

| | <ul> <li>Cosmética</li> <li>Acionada eletricamente</li> <li>Outra</li> </ul> |
|---|---|
| 5. | Que articulação repor a prótese |
| | <ul> <li>Ombro</li> <li>Cotovelo</li> <li>Pulso</li> <li>Dedos</li> </ul> |
| 6. | Que tão frequentemente usa sua prótese |
| | <ul> <li>Diário</li> <li>Ocasionalmente</li> <li>Nunca</li> </ul> |
| 7. | Qual área você acha que as prótese tem mais problemas |
| | <ul> <li>Encaixe da prótese</li> <li>Função</li> <li>Estética</li> <li>Mantenimento</li> <li>Peso do dispositivo</li> </ul> |
| 8. | Você usa a prótese em seu trabalho |
| 9. | <ul> <li>Sim</li> <li>Não</li> <li>Não trabalho</li> </ul> Usa a prótese para praticar esportes ou em atividades de lazer |
| | ■ Sim<br>■ Não |
| 10. | Quantas horas no dia aproximadamente usa a prótese: |
| 11. | Você dirige com o dispositivo ■ Sim ■ Não |
| 12. | Que tão satisfeito esta com seu dispositivo?: |
| 13. | Qual funcionalidade adicionaria em seu dispositivo?: |
| 14. | Quantas horas no dia aproximadamente usa a prótese: |
| 15. | O peso de seu dispositivo causa desconforto? |
| | ■ Sim<br>■ Não |
| 16. | Qual característica de seu dispositivo é a mais importante para você? |
| | 5 |





# 7.2. Questionário familiares

| 1. | Relação com o usuário |
|----|-------------------------------------------------------------------------|
| | ■ Esposa/Esposo |
| | ■ Pai/Mãe |
| | ■ Filho/Filha |
| | • Outro: |
| 2. | Idade |
| | ■ 18-20 |
| | <b>21-30</b> |
| | ■ 31-40 |
| | <b>4</b> 1-50 |
| | ■ 51-60 |
| | <b>+</b> 60 |
| 3. | Tipo de prótese que usa seu familiar |
| | ■ Cosmética |
| | ■ Acionada eletricamente |
| | ■ Outra |
| 4. | Qual área você acha que a prótese de seu familiar tem mais problemas |
| | ■ Encaixe da prótese |
| | ■ Função |
| | ■ Estética |
| | <ul> <li>Mantenimento</li> </ul> |
| | ■ Peso do dispositivo |
| 5. | Que tão satisfeitas acha que a pessoa esta com seu dispositivo?: |
| 6. | Qual área que você acha causa maior desconforto no uso do dispositivo?: |
| 7. | Qual funcionalidade adicionaria na prótese?: |
| 8. | Você acha que o peso da prótese dispositivo causa desconforto? |
| | ■ Sim |
| | ■ Não |
| 9. | Qual característica do dispositivo você acha é a mais importante? |





# 7.3. Questionário terapeutas

| 1. | Relação com o usuário |
|----|------------------------------------------------------------------------|
| 2. | Idade |
| | ■ 18-20 |
| | ■ 21-30 |
| | ■ 31-40 |
| | ■ 41-50 |
| | ■ 51-60 |
| | ■ +60 |
| 3. | Com qual tipo de próteses trabalha |
| | ■ Cosmética |
| | ■ Acionada eletricamente |
| | ■ Outra |
| 4. | Qual área você acha que as próteses que trabalha tem mais problemas |
| | ■ Encaixe da prótese |
| | ■ Função |
| | ■ Estética |
| | ■ Mantenimento |
| | ■ Peso do dispositivo |
| 5. | Que tão satisfeitas acha que as pessoas estão com seus dispositivos?: |
| 6. | Qual área que você acha causa maior desconforto no uso do dispositivo: |
| 7. | Qual funcionalidade adicionaria na prótese?: |
| 8. | Você acha que o peso da prótese dispositivo causa desconforto? |
| | ■ Sim |
| | ■ Não |
| 9. | Qual característica do dispositivo você acha é a mais importante? |